CLINICAL TRIAL: NCT00722098
Title: Melanoma Peptide-Loaded Dendritic Cell Vaccine in HLA-A*0201 Patients With Stage IV Melanoma: A Phase II Randomized Trial to Compare Vaccination With and Without Cyclophosphamide Treatment.
Brief Title: Comparison Study of Dendritic Cell Vaccine With and Without Cyclophosphamide to Treat Stage IV Melanoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to lesser accrual, and data analysis not done.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Baylor IRB #006-123
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Malignant Melanoma Stage IV
Keywords: Melanoma; Dendritic Cell; Vaccine; Immunotherapy; Cyclophosphamide
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DC Vaccine & Cyclophosphamide (Experimental): Patients will receive a fixed dose of about ≥15x106 viable dendritic cells per injection. Patients will receive a total of 8 doses of the vaccination with each individual dose being administered at weeks: 0, 2, 4, 6, 10, 14, 18 and 22. Responses will be evaluated and patients with SD, PR or CR may receive 4 more vaccine at 36, 48, 72 and 96 weeks, if there is vaccine available. The vaccine will be injected subcutaneously, in 3 separate injection sites (3.3.ml per site) in the upper and lower extremities.
  Patients will receive either CPA 300mg/m2 for injections administered intravenously over a 2-hour infusion in the outpatient clinic 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7.
  Interventions: Biological: DC Vaccine & Cyclophosphamide
- DC Vaccine & Placebo (Placebo Comparator): Patients will receive a fixed dose of about ≥15x106 viable dendritic cells per injection. Patients will receive a total of 8 doses of the vaccination with each individual dose being administered at weeks: 0, 2, 4, 6, 10, 14, 18 and 22. Responses will be evaluated and patients with SD, PR or CR may receive 4 more vaccine at 36, 48, 72 and 96 weeks, if there is vaccine available. The vaccine will be injected subcutaneously, in 3 separate injection sites (3.3.ml per site) in the upper and lower extremities.
  Patients will receive saline for injections administered intravenously over a 2-hour infusion in the outpatient clinic 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7.
  Interventions: Biological: DC Vaccine & Placebo

INTERVENTIONS:
Biological: DC Vaccine & Cyclophosphamide — Patients will receive a fixed dose of about ≥15x106 viable dendritic cells per injection. Patients will receive a total of 8 doses of the vaccination with each individual dose being administered at weeks: 0, 2, 4, 6, 10, 14, 18 and 22. Responses will be evaluated and patients with SD, PR or CR may receive 4 more vaccine at 36, 48, 72 and 96 weeks, if there is vaccine available. The vaccine will be injected subcutaneously, in 3 separate injection sites (3.3.ml per site) in the upper and lower extremities.
  Patients will receive either CPA 300mg/m2 for injections administered intravenously over a 2-hour infusion in the outpatient clinic 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7.
  Other Names: Cyclophosphamide (CPA); DC Vaccine ( Dendritic cell vaccine)
  Arms: DC Vaccine & Cyclophosphamide
Biological: DC Vaccine & Placebo — Patients will receive a fixed dose of about ≥15x106 viable dendritic cells per injection. Patients will receive a total of 8 doses of the vaccination with each individual dose being administered at weeks: 0, 2, 4, 6, 10, 14, 18 and 22. Responses will be evaluated and patients with SD, PR or CR may receive 4 more vaccine at 36, 48, 72 and 96 weeks, if there is vaccine available. The vaccine will be injected subcutaneously, in 3 separate injection sites (3.3.ml per site) in the upper and lower extremities.
  Patients will receive saline for injections administered intravenously over a 2-hour infusion in the outpatient clinic 24 hours prior to DC vaccinations # 1, 3, 5, 6 and 7.
  Other Names: DC Vaccine - Dendritic Cell Vaccine
  Arms: DC Vaccine & Placebo

SUMMARY:
The purpose of this study is to determine whether the combination of chemotherapy (Cyclophosphamide) and CD34-DC vaccines results in the improved rate of clinical responses for stage IV melanoma patients.

DETAILED DESCRIPTION:
Vaccination of patients with metastatic melanoma using ex vivo generated dendritic cells (DCs) loaded with tumor-associated antigen(s) have been shown to induce tumor-specific immunity against melanoma antigens measured by in vitro assays and, in some cases, tumor regression. At the present time, the numbers of recorded patients with metastatic melanoma who have been treated with DC vaccinations are too small to predict with certainty the future of overall therapeutic value of DC vaccinations in the management of patients with metastatic melanoma. The purpose of this study is to gather data on feasibility and efficacy of novel combination therapy of CPA and a DC vaccine outlined in this protocol to treat metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven metastatic melanoma, Stages M1a, M1b, M1c
2. HLA-A*0201 phenotype
3. Age: 21-75 years
4. ECOG performance status 0-1
5. Measurable metastatic melanoma lesions by physical examination or radiographs or scans.
6. Adequate marrow function:

   * White count ≥ 4,000/microliter: Subjects who have recently completed chemotherapy will be allowed study entry with White count ≥ 3,500/microliter
   * Hemoglobin ≥ 10.0 gm: Subjects who have recently completed chemotherapy will be allowed study entry with Hemoglobin ≥ 9.0 gm.
   * Platelets ≥ 100,000/microliter
7. Adequate hepatic function:

   * Bilirubin ≤ 1.5/mg/dL
   * Alkaline phosphatase ≤ 5 times the upper limit of normal
   * SGOT ≤ 5 times the upper limit of normal
   * SGPT ≤ 5 times the upper limit of normal
8. Adequate renal function:

   * Serum creatinine ≤ 1.5/mg/dL
9. No active CNS metastatic disease at screening.

   * Patients with a history of CNS melanoma lesions must have had lesions resected by surgery and/or gamma knife irradiation at least 3 months prior to study entry.
   * The total number of CNS lesions at diagnosis should not have exceeded 3.
10. Written informed consent

Exclusion Criteria:

1. Patients who have received > 8 cycles of cytotoxic chemotherapy or metastatic melanoma
2. Patients who have received any chemotherapy < 4 weeks before the beginning of the trial
3. Patients who have received interferon alpha (IFNα-2b) or sargramostim (GM-CSF) < 4 weeks before the beginning of the trial
4. Patients who have received high-dose interleukin-2 (IL-2) < 4 weeks before the beginning of the trial
5. Patients that have been diagnosed with more than 3 CNS melanoma lesions.
6. Patients that have been diagnosed with more than 5 hepatic metastases or any hepatic metastasis > 5 cm.
7. Baseline serum LDH > 1.1 times the upper limit of normal
8. Patients who are HIV+ (HIV patients are often profoundly immunodeficient because of the viral infection and this additional parameter will interfere with the evaluation of DC induced immune responses in melanoma patients. Furthermore, the safety of collecting DCs, loading them with antigen and re-infusing these cells to HIV+ patients has not yet been determined.)
9. Pregnancy (Pregnancy is associated with considerable immunosuppression 70 and this additional parameter will interfere with the evaluation of DC induced immune responses in melanoma patients. In addition, the safety and tolerability of cell body-loaded DC given subcutaneously is entirely unknown.)
10. Patients who have received corticosteroids or other immunosuppressive agents < 4 weeks before beginning the trial
11. Patients with active asthma and/or on treatment for asthma
12. Patients with angina pectoris
13. Patients with congestive heart failure
14. Patients with a history of autoimmune disease including lupus erythematosus, rheumatoid arthritis or thyroiditis
15. Patients with active infections including viral hepatitis
16. Patients with a history of neoplastic disease other than melanoma < 5 years prior to entry on the trial except for patients with carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin. Patients who have any of these two types of cancer and melanoma can be included.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Induction of melanoma-specific CD8+T Cell Immunity. | 2 years

SECONDARY OUTCOMES:
Rate of objective clinical responses. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fay, M.D., Principal Investigator — Baylor Institute for Immunology Research: Baylor University Medical Center
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States